CLINICAL TRIAL: NCT05342571
Title: Stress and Immunity in Lung Cancer Patients: Pilot Test of a Biobehavioral/Cognitive (ABC) Treatment for Stress, Depression, and Anxiety
Brief Title: A Biobehavioral/Cognitive Treatment for Stress, Depression, and Anxiety in Patients With Stage IV Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Barbara Andersen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-20339; NCI-2020-08120 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-11-29; First posted 2022-04-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Advanced Lung Carcinoma; Metastatic Lung Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (ABC session, surveys, biospecimen collection) (Experimental): Phase 1 of the intervention (10 weeks) will follow the following agenda: 1) Overview and progressive muscle relaxation, 2) Seeking and asking for disease-related and treatment-related information, 3) Problem solving skills, 4) Breathing techniques and sleep hygiene, 5) Assertive communication skills, 6) Identifying social network, 7) Asking for support, 8) Further information on social support, 9) Physical activity, and 10) Review of major topics, transition. Phase 2 of the intervention (4 weeks) which will be completed only by patients who do not experience remission in depressive symptoms by the end of phase 1, will follow the following agenda: 1) Identifying negative thoughts and problematic thinking patterns, 2) Generating alternative thoughts, 3) Behavioral activation, and 4) Review and wrap-up, transition to optional maintenance. Each session in Phase 1 and Phase 2 occurs once per week, for 60 minutes each. Maintenance sessions occur monthly, 60 minutes each.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Informational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Behavioral, Psychological or Informational Intervention — Participate in ABC session
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected
Other: Electronic Health Record Review — Medical records reviewed
Other: Informational Intervention — Receive patient guidebook
Other: Survey Administration — Complete surveys

SUMMARY:
This phase IIb trial studies the effect of a biobehavioral/cognitive (ABC) treatment on stress, depression, and anxiety in patients with stage IV lung cancer. Advanced lung cancer and stress or depression are associated with increased inflammation and decreased immunity. ABC is a combination of biobehavioral intervention, which studies the interaction between behavioral and biological processes, and cognitive therapy for the treatment for anxiety and depressive disorders. Giving ABC during lung cancer treatment may reduce stress, depression, and anxiety, and improve patients' quality of life and health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct a phase IIb pilot of a biobehavioral/cognitive (ABC) therapy intervention for patients with advanced (stage IV) lung cancer (N=40) with moderate to severe depressive symptoms and determine feasibility and treatment adherence.

II. Mode of delivery (in person, virtual), frequency of contact, and duration of contacts are studied to identify efficiencies to achieve clinical change.

SECONDARY OBJECTIVES:

I. Pre/post treatment change on patient reported outcomes (PROs) for depressive symptoms, anxiety symptoms, cancer specific stress, and physical symptoms.

II. Compare patients' ABC outcomes to responses of a matched sample (n=40) of patients previously accrued to BLCIO (Beating Lung Cancer in Ohio; ClinicalTrials.gov Identifier: NCT03199651) completing the same measures at equivalent time points using archival, deidentified data.

TERTIARY OBJECTIVES:

I. To evaluate effects of ABC on prognostic cell numbers/ratios (i.e., neutrophil/lymphocyte ratio, platelet/lymphocyte ratio, and advanced lung cancer inflammation indices) from patients pre to post ABC and comparable time points for the matched BLCIO sample using electronic medical record (eMR) data.

II. To evaluate effects of ABC on immunity, conducting correlative studies of inflammation, immune suppressive cells, and downstream effects on T- and natural killer (NK) cell function, using serum samples from ABC patients drawn at accrual, prior to cancer treatment, and 1 and 2 months during treatment.

OUTLINE:

INTENSIVE I PHASE: Patients participate in ABC sessions consisting of weekly, hour-long sessions for 10 weeks.

INTENSIVE II PHASE: Patients not achieving full remission after the first 10 weeks receive 4 additional weekly sessions.

MAINTENANCE PHASE (Optional): Patients may participate in 1 ABC session monthly for 4 months. These maintenance sessions serve as "booster" sessions.

Patients' medical records are reviewed, and will receive a patient guidebook to provide session-by-session descriptions to assist the patient to focus on the content and homework assignment completion. Patients also complete surveys at pre-treatment, every 2 months during cancer treatment, at post-treatment, and at 1 and 2 months follow-up. Patients also undergo blood collection at the time of initial diagnostic work-up, and at protocol weeks 5, 10, and 15.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with advanced (stage IV) lung cancer with diagnosis and staging confirmed by pathology report
* Moderate to severe symptoms of depression (>= 8 on Patients Health Questionaire-9) and/or moderate to severe symptoms of anxiety (>= 10 on Generalized Anxiety Disorder-7; GAD-7)
* English-speaking
* Willingness to provide access to medical records, provide biospecimens, and responses to patient reported outcome (PRO) assessments
* Ability to understand and willingness to sign an informed consent document

Exclusion Criteria:

* Patients to be treated with definitive chemo-radiotherapy
* Presence of untreated brain metastases
* Previous lung cancer diagnosis
* Presence of disabling hearing, vision, or impairing psychiatric conditions (e.g., psychosis, bipolar disorder, substance abuse) preventing consent or completion of self-report measures in English
* Imminent risk of suicide that precludes outpatient treatment
* Currently receiving psychological treatment/counseling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Acceptability, measured by Patient Satisfaction Survey (PSS) | Up to 2 months post-treatment
  Descriptive statistics of Patient Satisfaction Survey scores will examine if patient satisfaction scores for a biobehavioral/cognitive (ABC) treatment are "mostly satisfied." The PSS is a 15-item measure which asks patients to rate each ABC intervention component on a 4-point Likert scale ranging from 1 ("not helpful at all") to 4 ("very helpful). Items are summed and averaged. An average score of 3 or higher is considered to represent treatment satisfaction.
Retention | Baseline up to 2 months post-treatment
  Descriptive statistics of patient enrollment and retention rate for ABC will also be used. Patient enrollment will be measured by counting the number of patients who sign consent and enroll onto the trial. Retention will be measured by calculating the number of patients who complete 7 of 14 sessions (50%).
Change of depressive symptoms using Patient Health Questionnaire-9 (PHQ-9) | Baseline up to 2 months post-treatment
  Dependent-samples t-tests will examine feasibility by testing change of depressive symptoms via the PHQ-9 from pre- to post-treatment. The PHQ-9 scores can range from 0 to 27, with higher scores indicating more severe depression.
Change of anxiety symptoms using Generalized Anxiety Disorder Scale (GAD-7) | Baseline up to 2 months post-treatment
  Dependent-samples t-tests will examine feasibility by testing change of anxiety symptoms via the GAD-7 from pre- to post-treatment. The GAD-7 scores can range from 0 to 21, with higher scores indicating more severe anxiety.
Biospecimen analysis: Neutrophil/lymphocyte ratio (NLR) | Baseline to Week 15
  Neutrophil/lymphocyte ratio (NLR) will be calculated by collecting neutrophil count and lymphocyte count from laboratory tests, and dividing neutrophil by lymphocyte count to receive the ratio. This will be conducted at 4 time points: baseline, week 5, week 10, and week 15. Changes in NLR over time will be evaluated using longitudinal mixed models within a joint modeling framework.
Biospecimen analysis: Platelet/lymphocyte ratio (PLR) | Baseline to Week 15
  Platelet/lymphocyte ratio (PLR) will be calculated by collecting platelet count and lymphocyte count from laboratory tests, and dividing platelets by lymphocyte count to receive the ratio. This will be conducted at 4 time points: baseline, week 5, week 10, and week 15. Changes in PLR over time will be evaluated using longitudinal mixed models within a joint modeling framework.
Biospecimen analysis: Inflammation (Interleukin-6) | Baseline to Week 15
  Inflammation will be calculated by conducting the Interleukin-6 (IL-6) immunoassay on patient blood samples. This will be conducted at 4 time points: baseline, week 5, week 10, and week 15. Changes in NLR over time will be evaluated using longitudinal mixed models within a joint modeling framework.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Andersen, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu